CLINICAL TRIAL: NCT00615212
Title: A Single Center, Single Sequence, Open-Label, Repeat-Dose Study to Investigate the Effect of GSK376501 on Hepatic Cytochrome P450 Activity in Healthy Adult Subjects
Brief Title: Effect of GSK376501 on CYP450 Activity in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIX110825
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Healthy Subjects,; Cytochrome P450 isoenzymes,; Repeat Dose; GSK376501,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Midazolam; Rosiglitazone; Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Subjects receiving midazolam (Active Comparator): Eligible subjects will receive midazolam oral syrup with a dose of 5 milligrams on Day 1.
  Interventions: Drug: Midazolam
- Subjects receiving rosiglitazone (Active Comparator): Eligible subjects will receive rosiglitazone oral tablet with a dose of 4 milligrams on Day 2.
  Interventions: Drug: Rosiglitazone
- Subjects receiving flurbiprofen (Active Comparator): Eligible subjects will receive flurbiprofen oral tablet with a dose of 50 milligrams on Day
  Interventions: Drug: Flurbiprofen
- Subjects receiving GSK376501 (Experimental): Eligible subjects will receive GSK376501 oral tablet with a dose of 75 milligrams from Day 4 to Day 10.
  Interventions: Drug: GSK376501
- Subjects receiving GSK376501+ midazolam (Experimental): Eligible subjects will receive GSK376501 oral tablet with a dose of 75 milligrams along with midazolam oral tablet of 5 milligrams on Day 11.
  Interventions: Drug: GSK376501; Drug: Midazolam
- Subjects receiving GSK376501 + rosiglitazone (Experimental): Eligible subjects will receive GSK376501 oral tablet with a dose of 75 milligrams along with rosiglitazone oarl tablet of 4 milligrams on Day 12.
  Interventions: Drug: GSK376501; Drug: Rosiglitazone
- Subjects receiving GSK376501 + flurbiprofen (Experimental): Eligible subjects will receive GSK376501 oral tablet with a dose of 75 milligrams along with flurbiprofen oral tablet of 50 milligrams on Day 13.
  Interventions: Drug: GSK376501; Drug: Flurbiprofen

INTERVENTIONS:
Drug: GSK376501 — GSK376501 oral tablet will be available with dosing strengths of 75 milligrams administered once daily. Biconvex, It will be a round, white film-coated tablets with both plain sides and no identifying markings.
  Arms: Subjects receiving GSK376501; Subjects receiving GSK376501 + flurbiprofen; Subjects receiving GSK376501 + rosiglitazone; Subjects receiving GSK376501+ midazolam
Drug: Midazolam — Midazolam oral syrup will be available with a dose of 5 milligrams administered once daily. It will be a clear, red to purplish-red, cherry-flavored syrup.
  Arms: Subjects receiving GSK376501+ midazolam; Subjects receiving midazolam
Drug: Rosiglitazone — Rosiglitazone oral tablet will be available with dosing strengths of 4 milligrams administered once daily. It will be a orange colored tablet debossed with SB on one side and 4 on the other.
  Arms: Subjects receiving GSK376501 + rosiglitazone; Subjects receiving rosiglitazone
Drug: Flurbiprofen — Rosiglitazone oral tablet will be available with dosing strengths of 50 milligrams administered once daily. It will be a blue, oval, film coated tablet.
  Arms: Subjects receiving GSK376501 + flurbiprofen; Subjects receiving flurbiprofen

SUMMARY:
This study is meant to assess potential inhibitory effects of GSK376501 on CYP450 isoenzymes 3A4, 2C8, 2C9. subjects will receive probe compounds and systemic levels of these substrates will be compared pre and post dosing of GSK376501.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a qualified physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as: a. pre-menopausal females with a documented tubal ligation or hysterectomy; or b. postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Body weight ≥ 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Demonstrates an average QTc interval < 450 msec (or < 480 msec in subjects with bundle branch block), an average PR interval < 200 msec, and a QRS duration < 110msec (manual or machine read) at screening or baseline

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Previous exposure to GSK376501.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Demonstrates symptomatic or asymptomatic arrhythmia of any clinical significance during screening.
* The subject has a positive pre-study drug/alcohol screen and is unwilling to abstain from 72 hours prior to dose until follow-up. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urinary cotinine levels indicative of smoking or history or use of tobacco or nicotine-containing products within 6 months prior to screening.
* Has a history of alcohol abuse or dependence within 12 months prior to the study. Alcohol abuse is defined as an average consumption of greater than 7 drinks per week for women or greater than 14 drinks per week for men. One alcohol drink is defined as the equivalent of 12 g of alcohol as follows: 5 oz/150 ml wine, 12 oz (360 ml) beer or 1.5 oz (45 ml) of 80 proof distilled spirits.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort, kava, ephedra [ma huang], gingko biloba, DHEA, vohimbe, saw palmetto, ginseng, red yeast rice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and is unwilling to abstain from use of these medications until the last pharmacokinetic or pharmacodynamic sample has been collected, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Use of caffeine- or xanthine-containing products for 24 hours prior to dose until the last pharmacokinetic sample has been collected.
* Consumption of any food or any beverage containing (alcohol, grapefruit or
* grapefruit juice, apple or orange juice, Seville oranges, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats). from 7 days prior to the first dose of study medication.
* Use of acetaminophen within 48 hours of the first dose and is unable or unwilling to discontinue use of acetaminophen until the last pharmacokinetic sample has been collected.
* Use of aspirin, aspirin-containing compounds, salicylates or nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours days of the first dose and is unwilling to abstain from use of these medications until the last pharmacokinetic sample has been collected.
* Use of liquid antacids (e.g. Maalox, Mylanta, Amphogel, milk of magnesia) or chewable antacids (e.g. TUMS™) within 48 hours of the first dose and is unwilling to abstain from use of these medications until the last dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Alkaline phosphatase value higher than 1.5 times the upper limit of normal at screening or at baseline.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), direct (conjugated) bilirubin, or CPK values higher than 1.25 times upper limit of normal at screening or at baseline.
* Fasting triglyceride level > 400 mg/dL (4.52 mmol/L) at screening or at baseline. Triglyceride levels within a 10% margin above this level will be considered on a case-by-case basis.
* Donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of or current congestive heart failure (NYHA Class I-IV symptoms)
* History of thyroid dysfunction or an abnormal thyroid function test as assessed by TSH as screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2008-02-15 (Actual); Study Completion 2008-02-15 (Actual)

PRIMARY OUTCOMES:
drug plasma levels midazolam: | Days 1 & 11
drug plasma levels rosiglitazone: | Days 2 & 12
drug plasma levels flurbiprofen: | Days 3 & 13

SECONDARY OUTCOMES:
adverse reactions,changes in laboratory values,changes in vital signs, & ECG changes: | Days 1-13
drug plasma levels GSK376501: | Days 4-13
Safety and tolerability during dosing with GSK376501, alone and in combination with the various probe substrates. | Up to Day 24
Daily predose trough GSK376501 plasma concentrations when administered alone for 7 days (Days 4-13). | for 7 days (Days 4-13).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study DIX110825 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110825?search=study&study_ids=DIX110825#rs